CLINICAL TRIAL: NCT03936283
Title: Development and Testing of a Mobile-health (M-health) Intervention Tool to Help Overweight and Obese Women Achieve Appropriate Gestational Weight Gain
Brief Title: Study of a Randomized Intervention Designed to Increase Exercise in Pregnancy
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1278778-12
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Gestational Weight Gain
Keywords: lifestyle; intervention; body weight; pregnancy; Overweight; Obesity; Signs and Symptoms; Body weight changes
MeSH Terms: conditions — Gestational Weight Gain; Body Weight; Overweight; Obesity; Signs and Symptoms; Body Weight Changes | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Intervention — The goal of the intervention is to help women increase their minutes of moderate-to-vigorous physical activity and to increase their knowledge of the IOM gestational weight gain guidelines. The lifestyle intervention will be delivered through telephone counseling sessions with a study dietician trained in motivational interviewing techniques, as well as through technology-based tools, automated text messages and core lifestyle intervention sessions.
  Arms: Lifestyle Intervention

SUMMARY:
This project aims to determine whether a mobile-health (m-health) tool, accessible via smartphone or website, intervention for overweight and obese pregnant women improves physical activity, gestational weight gain, quality of life, stress and depression during pregnancy. This study will examine factors associated with using the m-health tool and the most highly utilized features of the tool, with a goal of understanding how it can be used and improved in future behavior change interventions. The hypothesis is that compared with usual care, an m-health intervention will result in increased minutes of moderate-to-vigorous physical activity and increased knowledge of the IOM GWG guidelines. The study design is a small pilot randomized trial to assess feasibility. This study will recruit and follow 70 overweight and obese pregnant women during the first trimester of pregnancy from Kaiser San Francisco and other facilities. The m-health intervention has the advantage of enabling overweight and obese women to monitor and improve their health behaviors without impacting the work flow of clinical care. Depending on the results of this initial evaluation, the clinical implications may include its implementation at the health system level and/or being evaluated and improved in the future by a larger investigation in a randomized controlled trial. The study team will assess adherence and acceptability of the intervention to inform future studies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Women aged 21 years or older receiving prenatal care at Kaiser Permanente San Francisco and Oakland and whose obstetric care clinicians approved their participation in the study;
* Pregravid BMI 25 to <40 (as determined from a measured pregravid weight in electronic medical record);
* Has access to a smartphone and Wi-Fi;
* Provides informed consent to participate.

Exclusion Criteria:

* Multiple births;
* Planning to move out of the area during the study period;
* Diagnosis of any of the following conditions: diabetes outside of pregnancy, severe disease of the cardio-pulmonary system, serious gastrointestinal disease (e.g., Crohn's disease, IBD), kidney disease, lung disease (e.g., emphysema, COPD), major psychiatric disorder, thyroid disease (diagnosed in the last month), cancer (not including non-malignant skin cancer), drug and alcohol abuse, or history of an eating disorder;
* History of bariatric surgery;
* Use of metformin or corticosteroids;
* Inability to speak, read, or understand English;
* Placed on bed rest at time of enrollment;
* >15 weeks' gestation at enrollment.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is only enrolling female participants.
Enrollment: 75 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Change in minutes of moderate physical activity as assessed by the Pregnancy Physical Activity Questionnaire (PPAQ) | Between 12 and 33 weeks of pregnancy
  The investigators will assess change in moderate to vigorous physical activity between surveys in pregnancy. The sports and exercise domain encompasses 20 PPAQ activities of moderate intensity (ranging 3 MET to 6 MET) and 2 PPAQ activities of vigorous intensity (6.5 MET and 7 MET). The volumes of all activities in the sports and exercise domain will be summed to arrive at an estimate of overall volume of moderate to vigorous intensity sports and exercise activity, expressed in MET hours per week. Higher levels of activity are generally associated with better outcomes. The distributions of all physical activity variables will be assessed for outliers.

SECONDARY OUTCOMES:
Increased knowledge of the current IOM gestational weight gain guidelines | Between 12 and 33 weeks of pregnancy
  Knowledge of the current IOM GWG guidelines (according to a woman's pre-pregnancy BMI) is assessed during two surveys in pregnancy. If the lower and upper bound provided by the patient are equivalent to or fall within the IOM recommendation bounds, then this will be classified as a match.

CONTACTS AND LOCATIONS:
Overall Officials: Monique M Hedderson, Ph.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas T, Xu F, Sridhar S, Sedgwick T, Nkemere L, Badon SE, Quesenberry C, Ferrara A, Mandel S, Brown SD, Hedderson M. A Web-Based mHealth Intervention With Telephone Support to Increase Physical Activity Among Pregnant Patients With Overweight or Obesity: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 Jun 22;6(6):e33929. doi: 10.2196/33929. PMID 35731565